CLINICAL TRIAL: NCT06733584
Title: Meeting the Needs of Young Hispanic Autistic Children: Developing a Culturally and Linguistically Sensitive Intervention to Alleviate Core Social Challenges
Brief Title: Meeting the Needs of Young Hispanic Autistic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Catholic Charities (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Pamela Rollins, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTD IRB-24-306; HT94252410184 / AR230003 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Autism
Keywords: Autism Intervention; Cultural and Linguistic Responsivity; Social development; Social communication; Hispanic
MeSH Terms: conditions — Autistic Disorder; Communication | interventions — Culture Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally and Linguistically Responsive Pathways with a Mutual Gaze Protocol (Experimental): 16 90-minute sessions (or 18 weeks, whichever comes first) of a Culturally and Linguistically Responsive adaptation of the Pathways manualized Naturalistic Developmental Behavioral Intervention (NDBI; research version). Pathways is parent-mediated and uses a coaching model.
  Interventions: Behavioral: Culturally and Linguistically Responsive Pathways Parent-Mediated Intervention
- Culturally and Linguistically Responsive Pathways without Mutual Gaze Protocol (Active Comparator): 16 90-minute sessions (or 18 weeks, whichever comes first) of a Culturally and Linguistically Responsive adaptation of the Pathways manualized Naturalistic Developmental Behavioral Intervention (NDBI; research version) without the Mutual Gaze Protocol. Pathways is parent-mediated and uses a coaching model.
  Interventions: Behavioral: Culturally and Linguistically Responsive Pathways Parent-Mediated Intervention without Mutual Gaze

INTERVENTIONS:
Behavioral: Culturally and Linguistically Responsive Pathways Parent-Mediated Intervention without Mutual Gaze — Pathways-trained bilingual research clinicians will conduct 90-minute weekly coaching sessions with caregivers in the family's home or other convenient location. Caregivers will receive a written and audio version of the program manual which has been adapted to be culturally and linguistically responsive to the Hispanic community. Sessions will review information about social communication, social sensory routines, and using naturalistic developmental behavioral strategies. Interventionists will demonstrate intervention strategies and provide caregivers with feedback and self-reflection.
  Arms: Culturally and Linguistically Responsive Pathways without Mutual Gaze Protocol
Behavioral: Culturally and Linguistically Responsive Pathways Parent-Mediated Intervention — Pathways-trained bilingual research clinicians will conduct 90-minute weekly coaching sessions with caregivers in the family's home or other convenient location. Caregivers will receive a written and audio version of the program manual which has been adapted to be culturally and linguistically responsive to the Hispanic community. Sessions will review information about social communication, infusing mutual gaze in social sensory routines, and using naturalistic developmental behavioral strategies. Interventionists will demonstrate intervention strategies and provide caregivers with feedback and self-reflection.
  Arms: Culturally and Linguistically Responsive Pathways with a Mutual Gaze Protocol

SUMMARY:
Purpose of the Study: The goal of this clinical trial is to find out if a technique called the "mutual gaze procedure" used in a Culturally and Linguistically Responsive adaptation of Pathways Early Intervention (CLR-Pathways) is the key to improving social communication, language, and everyday skills in young (18-42 months) Hispanic autistic children experiencing low income.

What Will Happen: Researchers will compare two versions of CLR-Pathways.

* Version 1: Includes mutual gaze strategies.
* Version 2: Does not include mutual gaze strategies.

What to Expect: Participants will:

* Attend 16 sessions (or 18 weeks if there are cancellations) of Pathways Intervention, each lasting 1.5 hours.
* Come to the clinic for a developmental check-up three times: before starting Pathways, right after completing Pathways, and three months after finishing Pathways.

DETAILED DESCRIPTION:
Study Description:

* Participants: 200 Hispanic autistic children experiencing low income and their caregivers will be randomly assigned to one of two groups in parallel:

  1. Group 1: CLR-Pathways Intervention with mutual gaze strategies.
  2. Group 2: CLR-Pathways Intervention without mutual gaze strategies.
* Intervention Sessions: Participants will attend 16 sessions, each lasting 1.5 hours, over approximately 18 weeks (allowing for possible cancellations) of parent-mediated intervention in their homes or another convenient location.

Assessments: To track progress and evaluate long-term effects, participants will undergo several culturally and linguistically appropriate assessments at three time points:

1. Baseline: Within two weeks before starting the intervention.
2. Post-Intervention: Within two weeks after completing the intervention.
3. Three-Month Follow-Up: 12-15 weeks after completing the intervention.

Each evaluation will take approximately 2-3 hours and will include:

* Child Assessments:

  * Autism Diagnostic Observation Schedule, Second Edition (ADOS-2; Lord et al., 2012): Researchers will use the ADOS-2 to assess communication, social interaction, play, and restricted/repetitive behaviors and to confirm a research diagnosis of autism (administered only at baseline)
  * Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4; Bayley & Aylward, 2019): Researchers will use the Bayley-4 to measure cognitive and motor skills (administered only at baseline)
  * Preschool Language Scales, Fifth Edition (PLS-5; Zimmerman et al., 2011): Researchers will use the English or Spanish version of the PLS-5 to assess receptive language age (administered only at baseline)
  * Communication and Symbolic Behavior Scales-Developmental Profile (CSBS-DP; Wetherby & Prizant, 2002): Researchers will use the CSBS-DP to evaluate social communication.
* Caregiver Questionnaires:

  * PhenX Toolkit Core Measures (PhenX; Hamilton et al., 2011): Researchers will use the PhenX to collect family and child demographic information, including parents' and grandparents' place of birth.
  * Vineland Adaptive Behavior Scales, Third Edition (VABS-III; Sparrow et al., 2016): Researchers will use the VABS-III to assess adaptive functioning.
  * Post-intervention Social Validity Questionnaire (Rollins et al., 2016): Researchers will use a questionnaire from a previous intervention efficacy study to assess the social validity of the intervention.

The CSBS-DP and VABS-III have been validated as appropriate measures for determining meaningful changes in children with or at high risk for autism, based on previous research.

• Video-Recorded Measures:

* Adult-Child Interactions (ACIs): Twelve-minute recordings will be transcribed and coded for social orienting, the Fluency and Connectedness and Joint Engagement measures of the Joint Engagement Rating Inventory (JERI; Adamson et al., 2020), intentional communication (EC Indicator; Greenwood et al., 2006), and expressive language.
* Parent-Child Interactions (PCIs): Twelve-minute naturalistic recordings will be coded for the Parent Calm Authority and Child Affiliative Obedience measures of the JERI.

ELIGIBILITY:
Inclusion Criteria:

* Children must be from a Hispanic family experiencing low income, defined as having an income-to-needs ratio of < 200% of the federal poverty level, determined by their household size
* Children must be between 18-42 months old at the start of the study
* Children must have no other known neurological or genetic concerns or disorders determined by parent report
* Children must receive a Calibrated Severity Score (CSS) of 4 or higher on the Autism Diagnostic Observational Schedule-2 (ADOS-2) administered by a qualified bilingual assessment associate
* Families must have a primary home language of English and/or Spanish

Exclusion Criteria:

* Children who are from a family that is not Hispanic and/or does not have an income-to-needs ratio of < 200% of the federal poverty level, determined by their household size
* Children younger than 18 months or older than 42 months at the start of the study
* Children whose parents report they have any other known neurological or genetic concerns or disorders
* Children who receive a Calibrated Severity Score (CSS) lower than 4 on the ADOS-2
* Families who do not have English or Spanish as a primary home language

Ages: 18 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Respeto | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Two dyadic measures of respeto will be coded using two items from the Joint Engagement Rating Inventory (JERI; Adamson et al., 2020). The Parent Calm Authority (PCA) subscale will measure the extent to which a parent influences the interaction using an assertive and confident yet gentle approach. The Child Affiliative Obedience (CAO) subscale will capture the child's affiliation, deference, and amenability to the parent's direction. These are scored using 7-point Likert scales (where 1 indicates no PCA or CAO, respectively). These measures will be derived from 12-minute naturalistic parent-child interaction video recordings. The interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked and subsequently coded for measures of respeto.
Change in Social Communication Skills | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Change in the raw scores obtained on the Social, Speech and Symbolic composites of The Communication and Symbolic Behavior Scales- Developmental Profile (CSBS-DP; Wetherby & Prizant, 2002) will be measured. Raw scores for the Social, Speech and Symbolic composites range from 0-64, 0-54 and 0-53 respectively (0 being the worst score). The CSBS-DP is a direct assessment of early social communication designed for children with a functional communication age between 6 months and 2 years.
Change in Adaptive Functioning | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Change in the raw scores obtained on the Communication, Daily Living, Socialization, and Motor Development domains of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II; Sparrow et al., 2005) will be measured. Raw scores for these domains range from 0-252, 0-286, 0-224, 0-154 respectively (lower scores being worse outcomes). The VABS-II is a standardized parent report measure of adaptive functioning designed for individuals from birth to age 90.
Change in Social Attention | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  The amount of time the child initiates eye gaze to the adult's eyes paired with positive affect will be measured (see Rollins et al., 2021 for a detailed description of this measure). This measure will be derived from 12-minute adult-child interaction video recordings wherein the child interacts with an unfamiliar adult during a semi-naturalistic play session. These interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked and subsequently coded for social orienting.
Change in Intentional Communication | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Intentional communication will be measured using the Early Communication Indicator (EC Indicator; Greenwood et al., 2006). The EC Indicator yields a total weighted communication score weighting gestures and vocalizations as 1, single words as 2 and multiple words as 3. Each utterance will also be coded for the child's attentional focus when communicating (attention to object, attention to adult, coordinated attention to object and adult). This measure will be derived from 12-minute adult-child interaction video recordings wherein the child interacts with an unfamiliar adult during a semi-naturalistic play session. These interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked, orthographically transcribed at the level of the utterance, and subsequently coded for intentional communication.
Change in Expressive Language | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Expressive language will be measured via the Moving Average Number of Different Words (MANDW) and Mean Length of Utterance in words (MLUw) calculated using the Systematic Analysis of Language Transcripts (SALT; Miller & Iglesias, 2020) software. MANDW measures expressive vocabulary using a moving window to estimate the number of different words, controlling for variability in length across language samples. MLUw measures combinatorial language by calculating the ratio of main body words to the number of utterances produced. This measure will be derived from 12-minute adult-child interaction video recordings wherein the child interacts with an unfamiliar adult during a semi-naturalistic play session. These interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked and orthographically transcribed.

SECONDARY OUTCOMES:
Change in Triadic Joint Attention | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Triadic joint attention will be measured using the Joint Engagement Rating Inventory (JERI; Adamson et al., 2020). Supported and Coordinated Joint Engagement subscales of the JERI will be used to capture the quantity and quality of the child paying active attention to both the parent and the shared object. They are scored using a 7-point Likert scale (with 1 indicating no episodes of supported or coordinated joint engagement, respectively). These measures will be derived from 12-minute adult-child interaction video recordings wherein the child interacts with an unfamiliar adult during a semi-naturalistic play session. These interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked and subsequently coded for triadic joint attention.
Change in Social Connectedness | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Social connectedness will be measured using the Fluency and Connectedness item of the Joint Engagement Rating Inventory (JERI; Adamson et al., 2020). Fluency and connectedness captures the flow of a dyad's interaction; it is scored using a 7-point Likert scale (with 1 indicating no episodes of coordinated joint engagement). This measure will be derived from 12-minute adult-child interaction video recordings wherein the child interacts with an unfamiliar adult during a semi-naturalistic play session. These interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked and subsequently coded for social connectedness.
Change in Proportion of Grammaticality | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Proportion of Grammaticality will be calculated using the Systematic Analysis of Language Transcripts (SALT; Miller & Iglesias, 2020) software. This captures the ability to conjugate verbs and use sentence structure grammatically. This measure will be derived from 12-minute adult-child interaction video recordings wherein the child interacts with an unfamiliar adult during a semi-naturalistic play session. These interactions will be video-recorded from a wide-angle view as well as from hidden camera eyeglasses worn by the adult to capture the location and direction of the child's eye gaze. The two streams of digitized videos will be time-linked and orthographically transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Rollins, EdD, Principal Investigator — The University of Texas at Dallas
Locations (3):
- United States (3):
  - University of Kansas, Lawrence, Kansas
  - Catholic Charities of Dallas, Dallas, Texas
  - University of Texas at Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
The shared data will include de-identified demographic data and item-level data from measures administered to participants, as well as analyzed data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data sharing schedule for demographic and study measure data is expected to begin approximately one year after the start of the project, with updates every 6 months. Analyzed data will be shared after the project is complete. It is our expectation that the data will persist in NDA's database for that organization's lifespan.
Access Criteria: The Database Engineer in the Research Design and Analysis (RDA) of the Life Span Institute at the KU will report the collected data to the National Institute of Mental Health Data Archive (NDA). NDA provides a robust system for defining data dictionaries and metadata for all datasets, and the uploaded data itself will be in delimited plain text format. Implementation of this data sharing plan will be the responsibility of RDA.

REFERENCES:
- [Background] Rollins PR, Campbell M, Hoffman RT, Self K. A community-based early intervention program for toddlers with autism spectrum disorders. Autism. 2016 Feb;20(2):219-32. doi: 10.1177/1362361315577217. Epub 2015 Apr 23. PMID 25907978
- [Background] Greenwood CR, Walker D, Buzhardt J, J Howard W, McCune L, Anderson R. Evidence of a Continuum in Foundational Expressive Communication Skills. Early Child Res Q. 2013 Jul 1;28(3):540-554. doi: 10.1016/j.ecresq.2013.02.006. PMID 24882940
- [Background] Hamilton CM, Strader LC, Pratt JG, Maiese D, Hendershot T, Kwok RK, Hammond JA, Huggins W, Jackman D, Pan H, Nettles DS, Beaty TH, Farrer LA, Kraft P, Marazita ML, Ordovas JM, Pato CN, Spitz MR, Wagener D, Williams M, Junkins HA, Harlan WR, Ramos EM, Haines J. The PhenX Toolkit: get the most from your measures. Am J Epidemiol. 2011 Aug 1;174(3):253-60. doi: 10.1093/aje/kwr193. Epub 2011 Jul 11. PMID 21749974
- [Background] Zimmerman, I. L., Steiner, V. G., & Pond, R. E. (2011). Preschool language scales (5th ed.). Pearson.
- [Background] Sparrow S. S., Cicchetti D. V., Balla D. A. (2005). Vineland Adaptive Behavior Scales, Second Edition (Vineland-II). San Antonio, TX: Pearson.
- [Background] Kosloski EE, Patel SD, Rollins PR. The Role of Pathways Early Autism Intervention in Improving Social Skills and Respeto for Young Hispanic Autistic Children. J Autism Dev Disord. 2025 Sep;55(9):3167-3178. doi: 10.1007/s10803-024-06419-x. Epub 2024 Jun 6. PMID 38842669
- [Background] Rollins PR, De Froy AM, Gajardo SA, Brantley S. Pragmatic contributions to early vocabulary and social communication in young autistic children with language and cognitive delays. J Commun Disord. 2022 Sep-Oct;99:106243. doi: 10.1016/j.jcomdis.2022.106243. Epub 2022 Jun 22. PMID 35797775
- [Background] Rollins PR, De Froy A, Campbell M, Hoffman RT. Mutual Gaze: An Active Ingredient for Social Development in Toddlers with ASD: A Randomized Control Trial. J Autism Dev Disord. 2021 Jun;51(6):1921-1938. doi: 10.1007/s10803-020-04672-4. PMID 32894382
- See also: This is the manual for the Joint Engagement Rating Inventory. [Adamson, L.B., Bakeman, R., & Suma, K. (2020). The joint engagement rating inventory. Department of Psychology, Georgia State University.] — https://sites.gsu.edu/bakeman/files/2024/03/DevLabTechReport25.4-397727a52df21a75.pdf
- See also: This is the link to the Autism Diagnostic Observation Schedule, Second Edition. [Lord, C., Luyster, R., Gotham, K., & Guthrie, W. (2012). Autism Diagnostic Observation Schedule (ADOS-2) (2nd ed.). Western Psychological Services.] — https://www.wpspublish.com/ados-2-autism-diagnostic-observation-schedule-second-edition
- See also: This is the link to the Bayley Scales of Infant and Toddler Development, Fourth Edition. [Bayley, N., & Aylward, G. P. (2019). Bayley Scales of Infant and Toddler Development (4th ed.). Pearson.] — https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Bayley-Scales-of-Infant-and-Toddler-Development-%7C-Fourth-Edition/p/100001996.html
- See also: This is a link to the Communication and Symbolic Behavior Scales. [Wetherby, A., & Prizant, B. (2002). Communication and Symbolic Behavior Scales- Developmental Profile (1st normed ed.). Paul H. Brookes.] — https://products.brookespublishing.com/Communication-and-Symbolic-Behavior-Scales-Developmental-Profile-CSBS-DP-First-Normed-Edition-P28.aspx